CLINICAL TRIAL: NCT05891405
Title: Cardiac Surgery for Babies Less Than 5 kg:Risk Factors for Morbidity and Mortality
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Atef Ahmed, Assistant lecturer, Sohag University
Other Study IDs: Soh-Med-23-05-02MD
Record Dates: First submitted 2023-05-28; First posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Cardiac Surgery in Neonates
MeSH Terms: interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cardiac surgery — Operations for congenital heart diseases

SUMMARY:
Cardiac surgery in babies less than 6 kg of weight is a complex and high-risk procedure. Despite advances in medical technology, mortality and morbidity rates remain high. This study seeks to identify risk factors associated with mortality and morbidity in this population

ELIGIBILITY:
Inclusion Criteria:

* neonates undergoing surgery for congenital heart diseases

Exclusion Criteria:

* larger body weights than 5 kg

Ages: 1 Day to 2 Years | Sex: All
Age Groups: Child
Study Population: Neonates with congenital heart diseases undergoing surgery for complete or partial treatment with body weight less than 5 kg at time of surgery
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | 1 month postoperative
  Death after surgery

SECONDARY OUTCOMES:
Morbidity | 1 month postoperative
  Complications after surgery